CLINICAL TRIAL: NCT00614575
Title: BI_Sifrol Tablets Special Drug Use Surveillance(Survey on the Safety and Efficacy in Parkinson's Disease Patients With Depressive Symptoms)
Brief Title: Survey on PD Patients With Depressive Symptoms
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Boehringer Ingelheim, Study Chair, Boehringer Ingelheim
Other Study IDs: 248.635
Record Dates: First submitted 2008-01-31; First posted 2008-02-13 (Estimated); Results first posted 2011-07-19 (Estimated); Last update posted 2014-08-06 (Estimated); Status verified 2014-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- BI-Sifrol® Tablets (Pramipexole): BI-Sifrol® Tablets, pramipexole dose: 0.125 mg, 0.5 mg, No reference therapy

SUMMARY:
The primary objective of this investigation is to conduct a 12-week prospective survey in PD patients with depressive symptoms treated with BI Sifrol Tablets (hereinafter referred to as this drug) in the routine clinical settings to determine the following items related to the safety and efficacy.

i. Adverse drug reaction symptoms, incidence, and severity ii. Motor capacity during the investigation iii. Depressive symptoms during the investigation

ELIGIBILITY:
Inclusion criteria:

**PD patients with depressive symptoms Patients who have not received pramipexole hydrochloride hydrate preparations within 1 month before survey entrance.

Exclusion criteria:

* PD patients with the past history of suicidal attempt, suicidal ideation or tendency
* PD patients with suicidal ideation
* PD patients with the past history of suicidal tendency

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: PD patients with depressive symptoms
Sampling Method: Non-Probability Sample
Enrollment: 1089 (Actual)
Dates: Start 2007-01; Primary Completion 2009-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (238):
- Japan (238):
  - Boehringer Ingelheim Investigational Site, Akashi
  - Boehringer Ingelheim Investigational Site 1, Akita
  - Boehringer Ingelheim Investigational Site 2, Akita
  - Boehringer Ingelheim Investigational Site, Asahikawa
  - Boehringer Ingelheim Investigational Site, Ashikaga
  - Boehringer Ingelheim Investigational Site, Awaji
  - Boehringer Ingelheim Investigational Site, Chitose
  - Boehringer Ingelheim Investigational Site, Chūō
  - Boehringer Ingelheim Investigational Site 1, Fuchū
  - Boehringer Ingelheim Investigational Site 2, Fuchū
  - Boehringer Ingelheim Investigational Site, Fuefuki
  - Boehringer Ingelheim Investigational Site, Fuehuki
  - Boehringer Ingelheim Investigational Site, Fujioka
  - Boehringer Ingelheim Investigational Site, Fujisaki
  - Boehringer Ingelheim Investigational Site, Fujisawa
  - Boehringer Ingelheim Investigational Site, Fukaya
  - Boehringer Ingelheim Investigational Site 1, Fukuoka
  - Boehringer Ingelheim Investigational Site 2, Fukuoka
  - Boehringer Ingelheim Investigational Site 3, Fukuoka
  - Boehringer Ingelheim Investigational Site 4, Fukuoka
  - Boehringer Ingelheim Investigational Site 5, Fukuoka
  - Boehringer Ingelheim Investigational Site 1, Fukushima
  - Boehringer Ingelheim Investigational Site 2, Fukushima
  - Boehringer Ingelheim Investigational Site, Funabashi
  - Boehringer Ingelheim Investigational Site 1, Gifu
  - Boehringer Ingelheim Investigational Site 2, Gifu
  - Boehringer Ingelheim Investigational Site, Habikino
  - Boehringer Ingelheim Investigational Site, Hachiōji
  - Boehringer Ingelheim Investigational Site 1, Hamamatsu
  - Boehringer Ingelheim Investigational Site 2, Hamamatsu
  - Boehringer Ingelheim Investigational Site 3, Hamamatsu
  - Boehringer Ingelheim Investigational Site 4, Hamamatsu
  - Boehringer Ingelheim Investigational Site 5, Hamamatsu
  - Boehringer Ingelheim Investigational Site, Hanamaki
  - Boehringer Ingelheim Investigational Site, Hayashima
  - Boehringer Ingelheim Investigational Site 1, Higashiosaka
  - Boehringer Ingelheim Investigational Site 2, Higashiosaka
  - Boehringer Ingelheim Investigational Site, Himeji
  - Boehringer Ingelheim Investigational Site, Hirakata
  - Boehringer Ingelheim Investigational Site, Hirishima
  - Boehringer Ingelheim Investigational Site, Hirosaki
  - Boehringer Ingelheim Investigational Site, Ibaraki
  - Boehringer Ingelheim Investigational Site, Iizuka
  - Boehringer Ingelheim Investigational Site, Inag
  - Boehringer Ingelheim Investigational Site, Irima
  - Boehringer Ingelheim Investigational Site, Isahaya
  - Boehringer Ingelheim Investigational Site, Iwaki
  - Boehringer Ingelheim Investigational Site, Iwamizawa
  - Boehringer Ingelheim Investigational Site, Iwata
  - Boehringer Ingelheim Investigational Site 1, Jyoetsu
  - Boehringer Ingelheim Investigational Site 2, Jyoetsu
  - Boehringer Ingelheim Investigational Site, Jyoyo
  - Boehringer Ingelheim Investigational Site 1, Kagoshima
  - Boehringer Ingelheim Investigational Site 2, Kagoshima
  - Boehringer Ingelheim Investigational Site 3, Kagoshima
  - Boehringer Ingelheim Investigational Site, Kahoku
  - Boehringer Ingelheim Investigational Site, Kamakura
  - Boehringer Ingelheim Investigational Site 1, Kanazawa
  - Boehringer Ingelheim Investigational Site 2, Kanazawa
  - Boehringer Ingelheim Investigational Site 1, Kanoya
  - Boehringer Ingelheim Investigational Site 2, Kanoya
  - Boehringer Ingelheim Investigational Site 1, Kashihara
  - Boehringer Ingelheim Investigational Site 2, Kashihara
  - Boehringer Ingelheim Investigational Site, Kasuga
  - Boehringer Ingelheim Investigational Site, Kawagchi
  - Boehringer Ingelheim Investigational Site, Kawaguchi
  - Boehringer Ingelheim Investigational Site 1, Kawasaki
  - Boehringer Ingelheim Investigational Site 2, Kawasaki
  - Boehringer Ingelheim Investigational Site, Kitakami
  - Boehringer Ingelheim Investigational Site 1, Kiyose
  - Boehringer Ingelheim Investigational Site 2, Kiyose
  - Boehringer Ingelheim Investigational Site, Kodaira
  - Boehringer Ingelheim Investigational Site, Kofu
  - Boehringer Ingelheim Investigational Site, Koga
  - Boehringer Ingelheim Investigational Site, Komae
  - Boehringer Ingelheim Investigational Site, Komatsu
  - Boehringer Ingelheim Investigational Site, Komatsushima
  - Boehringer Ingelheim Investigational Site, Koshigaya
  - Boehringer Ingelheim Investigational Site 1, Kōriyama
  - Boehringer Ingelheim Investigational Site 2, Kōriyama
  - Boehringer Ingelheim Investigational Site, Kōtari
  - Boehringer Ingelheim Investigational Site 1, Kumamoto
  - Boehringer Ingelheim Investigational Site 2, Kumamoto
  - Boehringer Ingelheim Investigational Site 3, Kumamoto
  - Boehringer Ingelheim Investigational Site, Kure
  - Boehringer Ingelheim Investigational Site, Kusatsu
  - Boehringer Ingelheim Investigational Site 1, Kyoto
  - Boehringer Ingelheim Investigational Site 2, Kyoto
  - Boehringer Ingelheim Investigational Site 3, Kyoto
  - Boehringer Ingelheim Investigational Site 4, Kyoto
  - Boehringer Ingelheim Investigational Site, Maebashi
  - Boehringer Ingelheim Investigational Site, Matsudo
  - Boehringer Ingelheim Investigational Site, Matsumoto
  - Boehringer Ingelheim Investigational Site, Mibu
  - Boehringer Ingelheim Investigational Site, Mihara
  - Boehringer Ingelheim Investigational Site, Mihoro
  - Boehringer Ingelheim Investigational Site, Miriyama
  - Boehringer Ingelheim Investigational Site, Misato
  - Boehringer Ingelheim Investigational Site, Miyako
  - Boehringer Ingelheim Investigational Site 1, Miyazaki
  - Boehringer Ingelheim Investigational Site 2, Miyazaki
  - Boehringer Ingelheim Investigational Site, Moriguchi
  - Boehringer Ingelheim Investigational Site 1, Morioka
  - Boehringer Ingelheim Investigational Site 2, Morioka
  - Boehringer Ingelheim Investigational Site, Moriya
  - Boehringer Ingelheim Investigational Site, Mukai-awagasaki
  - Boehringer Ingelheim Investigational Site, Musashino
  - Boehringer Ingelheim Investigational Site, Nagano
  - Boehringer Ingelheim Investigational Site, Nagaoka
  - Boehringer Ingelheim Investigational Site 1, Nagoya
  - Boehringer Ingelheim Investigational Site 2, Nagoya
  - Boehringer Ingelheim Investigational Site 3, Nagoya
  - Boehringer Ingelheim Investigational Site 4, Nagoya
  - Boehringer Ingelheim Investigational Site 1, Nara
  - Boehringer Ingelheim Investigational Site 2, Nara
  - Boehringer Ingelheim Investigational Site, Narashino
  - Boehringer Ingelheim Investigational Site, Narita
  - Boehringer Ingelheim Investigational Site, Narutō
  - Boehringer Ingelheim Investigational Site, Nasushiobara
  - Boehringer Ingelheim Investigational Site, Nichinan
  - Boehringer Ingelheim Investigational Site, Ninohe
  - Boehringer Ingelheim Investigational Site, Nishinomiya
  - Boehringer Ingelheim Investigational Site, Nishitōkyō
  - Boehringer Ingelheim Investigational Site, Okaya
  - Boehringer Ingelheim Investigational Site 1, Okayama
  - Boehringer Ingelheim Investigational Site 2, Okayama
  - Boehringer Ingelheim Investigational Site, Okazaki
  - Boehringer Ingelheim Investigational Site, Okinawa
  - Boehringer Ingelheim Investigational Site, Omuta
  - Boehringer Ingelheim Investigational Site 1, Osaka
  - Boehringer Ingelheim Investigational Site 2, Osaka
  - Boehringer Ingelheim Investigational Site 3, Osaka
  - Boehringer Ingelheim Investigational Site 4, Osaka
  - Boehringer Ingelheim Investigational Site 5, Osaka
  - Boehringer Ingelheim Investigational Site 6, Osaka
  - Boehringer Ingelheim Investigational Site, Ōgaki
  - Boehringer Ingelheim Investigational Site, Ōiso
  - Boehringer Ingelheim Investigational Site 1, Ōita
  - Boehringer Ingelheim Investigational Site 2, Ōita
  - Boehringer Ingelheim Investigational Site 3, Ōita
  - Boehringer Ingelheim Investigational Site, Ōmura
  - Boehringer Ingelheim Investigational Site, Ōnojō
  - Boehringer Ingelheim Investigational Site, Ōta-ku
  - Boehringer Ingelheim Investigational Site, Ōtake
  - Boehringer Ingelheim Investigational Site, Ōtsu
  - Boehringer Ingelheim Investigational Site, Ryūgasaki
  - Boehringer Ingelheim Investigational Site, Saeki
  - Boehringer Ingelheim Investigational Site, Saga
  - Boehringer Ingelheim Investigational Site 1, Sagamihara
  - Boehringer Ingelheim Investigational Site 2, Sagamihara
  - Boehringer Ingelheim Investigational Site 3, Sagamihara
  - Boehringer Ingelheim Investigational Site, Saijyo
  - Boehringer Ingelheim Investigational Site, Saitama
  - Boehringer Ingelheim Investigational Site 1, Sakai
  - Boehringer Ingelheim Investigational Site 2, Sakai
  - Boehringer Ingelheim Investigational Site 1, Sapporo
  - Boehringer Ingelheim Investigational Site 2, Sapporo
  - Boehringer Ingelheim Investigational Site 3, Sapporo
  - Boehringer Ingelheim Investigational Site 4, Sapporo
  - Boehringer Ingelheim Investigational Site 5, Sapporo
  - Boehringer Ingelheim Investigational Site 6, Sapporo
  - Boehringer Ingelheim Investigational Site 7, Sapporo
  - Boehringer Ingelheim Investigational Site 8, Sapporo
  - Boehringer Ingelheim Investigational Site 9, Sapporo
  - Boehringer Ingelheim Investigational Site, Sekigahara
  - Boehringer Ingelheim Investigational Site 1, Sendai
  - Boehringer Ingelheim Investigational Site 2, Sendai
  - Boehringer Ingelheim Investigational Site, Shimoda
  - Boehringer Ingelheim Investigational Site 1, Shimotsuke
  - Boehringer Ingelheim Investigational Site 2, Shimotsuke
  - Boehringer Ingelheim Investigational Site, Shinngu
  - Boehringer Ingelheim Investigational Site, Shiroishi
  - Boehringer Ingelheim Investigational Site 1, Shizuoka
  - Boehringer Ingelheim Investigational Site 2, Shizuoka
  - Boehringer Ingelheim Investigational Site, Shōwajima
  - Boehringer Ingelheim Investigational Site 1, Suita
  - Boehringer Ingelheim Investigational Site 2, Suita
  - Boehringer Ingelheim Investigational Site, Susono
  - Boehringer Ingelheim Investigational Site, Suzuka
  - Boehringer Ingelheim Investigational Site 1, Takaoka
  - Boehringer Ingelheim Investigational Site 2, Takaoka
  - Boehringer Ingelheim Investigational Site, Takatsuki
  - Boehringer Ingelheim Investigational Site, Tarimizu
  - Boehringer Ingelheim Investigational Site, Togitsu
  - Boehringer Ingelheim Investigational Site, Tokoname
  - Boehringer Ingelheim Investigational Site, Tokushima
  - Boehringer Ingelheim Investigational Site, Tokyo Arakawa-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Bunkyo-ku
  - Boehringer Ingelheim Investigational Site 1, Tokyo Chuo-ku
  - Boehringer Ingelheim Investigational Site 2, Tokyo Chuo-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Daito-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Koto-ku
  - Boehringer Ingelheim Investigational Site 1, Tokyo Meguro-ku
  - Boehringer Ingelheim Investigational Site 2, Tokyo Meguro-ku
  - Boehringer Ingelheim Investigational Site 1, Tokyo Minato-ku
  - Boehringer Ingelheim Investigational Site 2, Tokyo Minato-ku
  - Boehringer Ingelheim Investigational Site 3, Tokyo Minato-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Nakano-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Nerima-ku
  - Boehringer Ingelheim Investigational Site 1, Tokyo Ota-ku
  - Boehringer Ingelheim Investigational Site 2, Tokyo Ota-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Setagaya-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Setagaya
  - Boehringer Ingelheim Investigational Site, Tokyo Shibuya-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Shinagawa-ku
  - Boehringer Ingelheim Investigational Site 1, Tokyo Shinjyuku-ku
  - Boehringer Ingelheim Investigational Site 2, Tokyo Shinjyuku-ku
  - Boehringer Ingelheim Investigational Site 3, Tokyo Shinjyuku-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Sibuya-ku
  - Boehringer Ingelheim Investigational Site, Tokyo Toshima-ku
  - Boehringer Ingelheim Investigational Site, Tokyo-Edogawa-ku
  - Boehringer Ingelheim Investigational Site, Tokyo-Itabashi-ku
  - Boehringer Ingelheim Investigational Site, Toride
  - Boehringer Ingelheim Investigational Site, Tosu
  - Boehringer Ingelheim Investigational Site 1, Toyama
  - Boehringer Ingelheim Investigational Site 2, Toyama
  - Boehringer Ingelheim Investigational Site 3, Toyama
  - Boehringer Ingelheim Investigational Site, Toyohashi
  - Boehringer Ingelheim Investigational Site, Toyokawa
  - Boehringer Ingelheim Investigational Site, Toyonaka
  - Boehringer Ingelheim Investigational Site, Ube
  - Boehringer Ingelheim Investigational Site, Ueda
  - Boehringer Ingelheim Investigational Site, Ushiku
  - Boehringer Ingelheim Investigational Site 1, Utsunomiya
  - Boehringer Ingelheim Investigational Site 2, Utsunomiya
  - Boehringer Ingelheim Investigational Site, Wakayama
  - Boehringer Ingelheim Investigational Site 1, Yachiyo
  - Boehringer Ingelheim Investigational Site 2, Yachiyo
  - Boehringer Ingelheim Investigational Site 3, Yachiyo
  - Boehringer Ingelheim Investigational Site, Yamanashi
  - Boehringer Ingelheim Investigational Site, Yanago
  - Boehringer Ingelheim Investigational Site, Yoichi
  - Boehringer Ingelheim Investigational Site 1, Yokohama
  - Boehringer Ingelheim Investigational Site 2, Yokohama
  - Boehringer Ingelheim Investigational Site 3, Yokohama
  - Boehringer Ingelheim Investigational Site 4, Yokohama
  - Boehringer Ingelheim Investigational Site, Yokosuka
  - Boehringer Ingelheim Investigational Site, Yoshinogawa

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The number of patients enrolled was 1089. The number of case reports collected from the patients enrolled in this survey was 1071. Moreover the number of patients analyzed as safety analysis was 1044, because 27 patients were excluded due to protocol violations.
Groups:
- BI-Sifrol Tablets: According to the dosage and administration described in the package insert of the drug in Japan, the drug was administered orally to PD patients with depressive symptoms under condition of routine medical practice. The description is as follows; Usually in adults, the starting dosage of pramipexole hydrochloride hydrate is 0.25 mg/day, followed by 0.5 mg/day during Week 2 of treatment, and the dosage is then increased by 0.5 mg/day each week under close observation to determine the maintenance dose (standard daily dose, 1.5-4.5 mg). When the daily dose of pramipexole hydrochloride hydrate is less than 1.5 mg, the daily dose will be divided into two doses to be taken after breakfast and after dinner. When the daily dose is 1.5 mg or higher, the daily dose will be divided into three doses to be taken after every meal. The dosage may be adjusted according to age and symptoms of the patient, but the daily dose should not exceed 4.5 mg.
Period: Overall Study
Arm/Group | BI-Sifrol Tablets
Started | 1089 (The number of patients enrolled.)
Completed | 861
Not Completed | 228
Not completed — Adverse Event | 106
Not completed — Lost to Follow-up | 55
Not completed — Lack of Efficacy | 14
Not completed — Withdrawal by Subject | 6
Not completed — Death | 3
Not completed — Physician Decision | 2
Not completed — No data were collected. | 18
Not completed — Irregularly enrolled patients | 23
Not completed — No treatment | 1

BASELINE CHARACTERISTICS:
Arm/Group | BI-Sifrol Tablets
Number analyzed (Participants) | 1044
Age, Continuous [Mean (Standard Deviation); unit: years] — The number of patients enrolled was 1089. The number of case reports collected from the patients enrolled in this survey was 1071. Moreover the number of patients analyzed as safety analysis was 1044, because 27 patients were excluded due to protocol violations.
  years | 70.5 (8.6)
Sex: Female, Male [Count of Participants; unit: Participants] — The number of patients enrolled was 1089. The number of case reports collected from the patients enrolled in this survey was 1071. Moreover the number of patients analyzed as safety analysis was 1044, because 27 patients were excluded due to protocol violations.
  Participants
    Female | 668
    Male | 376

OUTCOME MEASURES:

1. Secondary Outcome: Clinical Global Impression of Improvement
Description: Investigators evaluation of the Parkinson's disease (PD) symptoms on the Clinical Global Impression (CGI) with 5 categories (very much improved, much improved, minimally improved, no effect, and unassessable).
Time Frame: for 12 weeks after initiation of the treatment
Population: Efficacy analysis set
Measure: Number; unit: participants
Arm/Group | BI-Sifrol Tablets
Number analyzed (Participants) | 949
participants
  Very much improved | 76
  Much improved | 399
  Minimally improved | 348
  No effect | 102
  Unassessable | 24

2. Secondary Outcome: Mean Change From Baseline in Unified Parkinson's Disease Rating Scale (UPDRS) Part III Total Score
Description: Part III of the UPDRS contains the clinician-scored motor evaluation, and includes 14 individual items each scored from 0 (Normal) to 4 (Extreme dysfunction). The total score ranged from 0 to 56. A negative change in the Part III total score indicates improvement.
Time Frame: Baseline and after 12 weeks (or at the time of discontinuation)
Population: Efficacy analysis set
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | BI-Sifrol Tablets
Number analyzed (Participants) | 933
Unit on a scale | -7.2 (9.0)
Statistical Analysis 1: Comparison: BI-Sifrol Tablets; Test type: Superiority or Other; p < 0.0001, Paired t-test; Mean change from baseline = -7.2, Standard Deviation 9.0

3. Secondary Outcome: Mean Change From Baseline in Beck's Depression Inventory (BDI) Total Score
Description: The degree of severity in depressive state are scored between 0-63 in BDI. A decrease in the score means improvement.
Time Frame: Baseline and after 12 weeks (or at the time of discontinuation)
Population: Efficacy analysis set
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | BI-Sifrol Tablets
Number analyzed (Participants) | 887
Unit on a scale | -4.8 (7.8)
Statistical Analysis 1: Comparison: BI-Sifrol Tablets; Test type: Superiority or Other; p < 0.0001, Paired t-test; Mean change from baseline = -4.8, Standard Deviation 7.8

4. Secondary Outcome: Mean Change From Baseline in UPDRS (Unified Parkinson's Disease Rating Scale) Part I Item 3 Score
Description: Unified Parkinson's Disease Rating Scale Part I Item 3 assesses the participant for symptoms of depression. Item 3 scores range from 0 (None) to 4 (Sustained depression with suicidal thoughts or intent). A higher score indicates more severe depression symptoms. A negative change in the item 3 score indicates improvement.
Time Frame: Baseline and after 12 weeks (or at the time of discontinuation)
Population: Efficacy analysis set
Measure: Mean (Standard Deviation); unit: Unit on a scale
Arm/Group | BI-Sifrol Tablets
Number analyzed (Participants) | 945
Unit on a scale | -0.7 (0.9)
Statistical Analysis 1: Comparison: BI-Sifrol Tablets; Test type: Superiority or Other; p < 0.0001, paired t-test; Mean change from baseline = -0.7, Standard Deviation 0.9

5. Secondary Outcome: Mean Change From Baseline in Modified Hoehn & Yahr Rating Scale
Description: This scale is an investigator-completed assessment of the degree of complications arising from Parkinson's disease. The scale ranges from 0 (No signs) to 5 (Bedridden). A negative change in the Yahr rating scale indicates improvement.
Time Frame: After 12 weeks or at the time of discontinuation
Population: Efficacy Analysis Set
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | BI-Sifrol Tablets
Number analyzed (Participants) | 945
units on a scale | -0.3 (0.6)
Statistical Analysis 1: Comparison: BI-Sifrol Tablets; Test type: Superiority or Other; p < 0.0001, paired t-test; mean change from baseline = -0.3, Standard Deviation 0.6

6. Primary Outcome: Percentage of Participants With Adverse Events, Adverse Drug Reactions, and Serious Adverse Events
Description: The aim of this Post Marketing Surveillance (PMS) was to obtain safety data with treatment of pramipexole in Parkinson's disease patients with depressive symptoms. The percentage of participants with adverse events, adverse drug reactions, and serious adverse events are presented.
Time Frame: for 12 weeks
Population: Safety Analysis Set
Measure: Number; unit: percentage of participants
Arm/Group | BI-Sifrol Tablets
Number analyzed (Participants) | 1044
percentage of participants
  Proportion of Adverse Events | 21.7
  Proportion of Adverse Drug Reactions | 19.2
  Proportion of Serious Adverse Events | 2.5

ADVERSE EVENTS:
Time Frame: 12 weeks
Description: Interview at each visit. The number of patients enrolled was 1089. The number of case reports collected from the patients enrolled in this survey was 1071. Moreover the number of patients analyzed as safety analysis was 1044, because 27 patients were excluded due to protocol violations.
Arm/Group | BI-Sifrol Tablets
Serious Adverse Events (participants affected / at risk) | 26/1044
Other Adverse Events (participants affected / at risk) | 71/1044
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BI-Sifrol Tablets (N=1044)
Bronchitis (Infections and infestations) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2)
Nasal sinus cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Large intestine carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Gastrointestinal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1)
Dehydration (Metabolism and nutrition disorders) | 1 (1)
Confusional state (Psychiatric disorders) | 1 (1)
Delirium (Psychiatric disorders) | 2 (2)
Delusion (Psychiatric disorders) | 3 (3)
Hallucination (Psychiatric disorders) | 4 (4)
Somatoform disorder (Psychiatric disorders) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1)
Dizziness (Nervous system disorders) | 1 (1)
Neuroleptic malignant syndrome (Nervous system disorders) | 1 (1)
Dementia with Lewy bodies (Nervous system disorders) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Dyspepsia (Gastrointestinal disorders) | 1 (1)
Gastric ulcer haemorrhage (Gastrointestinal disorders) | 1 (1)
Ileus (Gastrointestinal disorders) | 1 (1)
Vomiting (Gastrointestinal disorders) | 1 (1)
Cholecystitis (Hepatobiliary disorders) | 1 (1)
Back pain (Musculoskeletal and connective tissue disorders) | 1 (1)
Prostatitis (Reproductive system and breast disorders) | 1 (1)
Death (General disorders) | 2 (2)
Fall (Injury, poisoning and procedural complications) | 3 (3)
Femoral neck fracture (Injury, poisoning and procedural complications) | 2 (2)
Fracture (Injury, poisoning and procedural complications) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | BI-Sifrol Tablets (N=1044)
Somnolence (Nervous system disorders) | 71 (71)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Any publication of the result of this trial must be consistent with the Boehringer Ingelheim publication policy. The rights of the investigator and of the sponsor with regard to publication of the results of this trial are described in the investigator contract.